CLINICAL TRIAL: NCT02047903
Title: An Observational Study of GIOTRIF (Afatinib) for First Line Therapy in Patients With Advanced Non Small Cell Lung Cancer (NSCLC) Harboring Epidermal Growth Factor Receptor (EGFR)-Mutations.
Brief Title: GIOTRIF in First Line Therapy of Advanced NSCLC With EGFR-mutations
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200.205
Record Dates: First submitted 2014-01-27; First posted 2014-01-28 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Afatinib
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — 50, 40, 30 or 20 mg

SUMMARY:
This observational study will investigate the efficacy, safety, tolerability and symptom control of GIOTRIF (Afatinib) in daily routine first-line therapy in patients with locally advanced or metastatic NSCLC harboring EGFR-mutations. Eligible NSCLC patients, for whom the treating physician has decided to initiate treatment with GIOTRIF in first line according to the local label, will be followed up for approximately 24 months.

DETAILED DESCRIPTION:
Study Design:

ELIGIBILITY:
Inclusion criteria:

* EGFR- tyrosine kinase inhibitor (TKI) naive patients with histologically confirmed locally advanced or metastatic NSCLC with activating EGFR-mutations
* Age >= 18 years
* No diagnostic or therapeutic measures beyond routine clinical practice are required
* Patients for whom the treating physician has decided to initiate treatment with GIOTRIF
* Written informed consent prior inclusion

Exclusion criteria:

* Contraindication for Afatinib according to the Summary of Product characteristics
* Participation in another clinical study until 30 days after end of treatment
* Prior systemic chemotherapy (Neo-/adjuvant therapy is permitted)
* Previous treatment with an EGFR-tyrosine kinase inhibitor
* Patients not willing or not able to fill in quality of life questionnaires
* Patients with missing or impaired legal capacity
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC-EGFR mutation positive
Sampling Method: Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2014-03-05 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Multiple Locations, Germany

REFERENCES:
- [Derived] Brueckl WM, Reck M, Schafer H, Neben K, Griesinger F, Rawluk J, Kruger S, Kokowski K, Ficker JH, Moller M, Schueler A, Laack E. Older patients with EGFR mutation-positive non-small cell lung cancer treated with afatinib in clinical practice: A subset analysis of the non-interventional GIDEON study. J Geriatr Oncol. 2023 Jan;14(1):101394. doi: 10.1016/j.jgo.2022.10.009. Epub 2022 Oct 30. PMID 36323612

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a non-interventional study (NIS) in real life clinical setting, in which responses were determined by using Response Evaluation Criteria in Solid Tumors (RECIST)/World Health Organization (WHO)/clinical evidence as investigators deemed appropriate.
Pre-assignment Details: Data source for this study were medical records usually collected during routine clinical practice other than study-specific questionnaires. Data collection was performed between March 24, 2014 and March 14, 2019.
Groups:
- Afatinib: Participants with locally advanced and /or metastatic non-small cell lung cancer (NSCLC) with activating epidermal growth factor receptor (EGFR) mutations received orally 40 milligram (mg) or less than 40 mg Afatinib starting dose once daily as first-line therapy. With dose escalation to maximum of 50 mg/day and reduction to 30 mg/day or 20 mg/day according to the summary of product characteristics (SmPC) under routine clinical conditions. The dose should not be escalated in any participant with a prior dose reduction.
Period: Overall Study
Arm/Group | Afatinib
Started | 161
Treated | 152
Completed | 102
Not Completed | 59
Not completed — Adverse Event | 14
Not completed — Serious adverse event | 10
Not completed — Withdrawal by Subject | 16
Not completed — Lost to Follow-up | 4
Not completed — Reason not listed | 6
Not completed — Not Treated | 9

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This patient set included all patients who received at least one dose of afatinib.
Arm/Group | Afatinib
Number analyzed (Participants) | 152
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.32 (10.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Rate After 12 Months
Description: The rate (probability) of being progression free after 12 months. PFS is defined as the time from first administration of the trial drug until objective tumor progression or death. The rate is the Kaplan-Meier estimated percent probability.
Time Frame: After 12 months
Population: Per protocol set (PPS): This set included all patients who gave their informed consent, did not violate any inclusion or exclusion criterion and have at least one documented administration of afatinib.
Measure: Number (95% Confidence Interval); unit: Percent probability of PFS
Arm/Group | Afatinib
Number analyzed (Participants) | 146
Percent probability of PFS | 50.24 [41.55 to 58.29]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate is calculated as a percentage of participants with complete response (CR) or partial response (PR) (i.e CR+PR) as best unconfirmed response. Here CR and PR were determined by investigators by using RECIST/WHO/clinical evidence as investigators deemed appropriate.
Time Frame: From the initial dose of study drug until end of the treatment period, up to 48 months.
Population: PPS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib
Number analyzed (Participants) | 146
Percentage of participants | 74.58 [65.74 to 82.14]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Percentage of participants with controlled disease (CR + PR + stable disease (SD)) as best unconfirmed response. CR, PR and SD were determined by investigators by using RECIST/WHO/clinical evidence as investigators deemed appropriate
Time Frame: From the initial dose of study drug until end of the treatment period, up to 48 months.
Population: PPS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib
Number analyzed (Participants) | 146
Percentage of participants | 91.53 [84.97 to 95.86]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was measured from start of therapy until progression or death, whichever came first. Progression was defined as the minimum of the first examination with progression and the date of progression documented by the treating physician. One day was added to the corresponding date. Patients without documented progression and not known to have died were censored at their date of last examination and one day was added. Median was derived by Kaplan Meier methods.
Time Frame: From first administration of the trial drug until objective tumour progression or death, up to 48 months.
Population: PPS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib
Number analyzed (Participants) | 146
Months | 12.17 [10.46 to 15.99]

5. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Percentage of participants with treatment emergent adverse events (TEAEs) and serious adverse events (SAEs).
Time Frame: From first administration of the trial drug until 30 days end after permanent discontinuation of therapy or end of study, up to 48 months.
Population: Treated set (TS): This patient set included all patients who received at least one dose of afatinib.
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib
Number analyzed (Participants) | 152
Percentage of participants
  AEs | 96.05
  SAEs | 42.76

6. Secondary Outcome: Toxicity and Side-effect Profile: Incidence of Diarrhea, Skin Reactions, Stomatitis and Paronychia
Description: Toxicity and side-effect profile: incidence of diarrhea, skin reactions, stomatitis and paronychia. Skin reactions: acne, dermatitis acneiform, dry skin, pruritus, rash, rash maculo-papular, rash pustular.
Time Frame: as for outcome 5
Population: TS
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib
Number analyzed (Participants) | 152
Percentage of participants
  Diarrhea | 82.89
  Stomatitis | 18.42
  Paronychia | 25.66
  Dermatitis acneiform | 37.50
  Acne | 1.32
  Dry skin | 16.45
  Pruritus | 10.53
  Rash | 5.26
  Rash maculo-papular | 17.76
  Rash pustular | 6.58

7. Secondary Outcome: Treatment Duration
Description: Duration of treatment with afatinib is calculated as Date of last administration + 1 day - Date of first administration.
Time Frame: From the initial dose of study drug until end of the treatment period, up to 48 months.
Population: TS
Measure: Median (Full Range); unit: Days
Arm/Group | Afatinib
Number analyzed (Participants) | 152
Days | 324.5 [13.0 to 1460.0]

8. Secondary Outcome: Symptom Control - Time to Worsening (Cough, Dyspnea and Pain)
Description: Symptom control was evaluated for cough, dyspnea and pain. Time to deterioration was calculated from date of baseline European Organisation for Research and Treatment of Cancer (EORTC) questionnaire until date of the EORTC questionnaire, where the first deterioration was measured. Patients without deterioration were censored at their date of last answered EORTC questionnaire, where the corresponding scale is evaluable. Participants had to select one answer on a scale ranging from 1=Not at All to 4=Very Much for questions 1 to 28 and 31 to 43 and on scale ranging from 1=Very Bad to 7=Excellent for questions 29 and 30. Afterwards, these scale scores were linearly transformed such that all scales ranged from 0 to 100, where higher scores represented higher level of symptoms.
Time Frame: Up to 48 months
Population: TS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib
Number analyzed (Participants) | 152
Months
  Cough: number analyzed (Participants) | 119
  Cough | 33.85 [17.86 to NA] — The upper limit was not reached
  Dyspnea: number analyzed (Participants) | 118
  Dyspnea | 22.17 [13.68 to NA] — The upper limit was not reached
  Pain: number analyzed (Participants) | 119
  Pain | 18.26 [9.21 to 23.72]

9. Secondary Outcome: Percentage of Participants With Treatment Modification
Description: Percentage of participants with treatment modification was calculated as percentage of participants with any dose reduction, dose escalation or any modification.
Time Frame: From the initial dose of study drug until end of the treatment period, up to 48 months.
Population: TS
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib
Number analyzed (Participants) | 152
Percentage of participants
  Any dose reduction | 59.87
  Dose increase | 17.11
  Any dose modifications | 61.84

ADVERSE EVENTS:
Time Frame: From first administration of the trial drug until 30 days end after permanent discontinuation of therapy or end of study, up to 48 months.
Arm/Group | Afatinib
All-Cause Mortality (participants affected / at risk) | 73/152
Serious Adverse Events (participants affected / at risk) | 65/152
Other Adverse Events (participants affected / at risk) | 144/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (N=152)
Anaemia (Blood and lymphatic system disorders) | 2
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Mitral valve disease (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Cataract (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Anal haemorrhage (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 22
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Pancreatitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Chest pain (General disorders) | 1
Death (General disorders) | 2
General physical health deterioration (General disorders) | 3
Pyrexia (General disorders) | 2
Pneumobilia (Hepatobiliary disorders) | 1
Arthritis infective (Infections and infestations) | 1
Biliary tract infection (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 4
Osteomyelitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Amylase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Lipase increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Renal colic (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Spinal operation (Surgical and medical procedures) | 1
Embolism (Vascular disorders) | 5
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (N=152)
Abdominal pain (Gastrointestinal disorders) | 12
Diarrhea (Gastrointestinal disorders) | 123
Nausea (Gastrointestinal disorders) | 20
Stomatitis (Gastrointestinal disorders) | 28
Vomiting (Gastrointestinal disorders) | 13
Fatigue (General disorders) | 23
Influenza like illness (General disorders) | 8
Nail infection (Infections and infestations) | 10
Paronychia (Infections and infestations) | 42
Rash pustular (Infections and infestations) | 10
Weight decreased (Investigations) | 9
Decreased appetite (Metabolism and nutrition disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 24
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 58
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 28
Pruritus (Skin and subcutaneous tissue disorders) | 16
Rash (Skin and subcutaneous tissue disorders) | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 27
Skin fissures (Skin and subcutaneous tissue disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT02047903/SAP_000.pdf
  • Study Protocol (2014-07-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT02047903/Prot_001.pdf